CLINICAL TRIAL: NCT03874949
Title: Comparison of Postoperative Pain After Root Canal Obturation With Sealer Containing or Not 1% Enoxolone: a Randomized Clinical Trial
Brief Title: Pain After Root Canal Obturation With Sealer Containing or Not 1% Enoxolone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACTEON Group (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEAU
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Root Canal Obturation

STUDY DESIGN:
Intervention Model Description: Subject will be randomized in a 1:1 allocation ratio between the two treatment groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEALITE Regular (Active Comparator): zinc oxide eugenol sealer
  Interventions: Device: SEALITE Regular
- SEALITE Ultra (Experimental): zinc oxide eugenol sealer containing 1% Enoxolone (NSAID)
  Interventions: Device: SEALITE Ultra

INTERVENTIONS:
Device: SEALITE Regular — Patients are treated with SEALITE Regular sealer (zinc oxide eugenol sealer). The SEALITE Regular powder is mixed with SEALITE Liquid according to the manufacturer instructions and added to gutta percha in the root canal for permanent obturation. The apical obturation is assessed by a postoperative radiographic control.
  Arms: SEALITE Regular
Device: SEALITE Ultra — Patients are treated with SEALITE Ultra sealer (zinc oxide eugenol sealer containing 1% Enoxolone).
  The SEALITE Ultra powder is mixed with SEALITE Liquid according to the manufacturer instructions and added to gutta percha in the root canal for permanent obturation. The apical obturation is assessed by a postoperative radiographic control.
  Arms: SEALITE Ultra

SUMMARY:
This study aims to assess the efficacy of a zinc oxide eugenol sealer containing Enoxolone, a non-steroidal anti inflammatory drug (NSAID) on the pain relief after endodontic treatment.

The study design is a multicenter, doubled blinded randomized controlled trial. The comparator is the equivalent zinc oxide eugenol sealer without NSAID (allocation ratio is 1:1). The conventional endodontic treatment, using gutta percha and sealer, is done. Patients assess their pain for 7 days after permanent root obturation.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged from 18 to 70 years,
* patient requiring root canal treatment on permanent mature teeth (single rooted teeth, premolar or molar),
* Informed consent signed,
* Patient with social protection.

Exclusion Criteria:

* root canal retreatment,
* root canal treatment on an immature tooth,
* calcified root canal assessed radiographically,
* Patient with one or more documented contraindication to endodontic treatment,
* Patient who takes regular analgesic or anti-inflammatory therapy for another pathology,
* Known allergy to NSAID or to one component of the sealer formula,
* Participation to another clinical trial at the same time,
* known pregnancy or lactation,
* Patients with legal protection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  To assess the efficacy of Enoxolone contained in the SEALITE Ultra formula compared to the SEALITE Regular formula, the pain is assessed by patients on a diary using a Visual Analogue Scale (VAS : 0-100 mm) 24 hours after the root canal obturation.

SECONDARY OUTCOMES:
Pain response profil | 0 hour, 6 hours, 12 hours, 24 hours, Day 2, Day 3, Day 7
  Patients reporte their pain in a diary at different times after endodontic treatment using a VAS : T0 (at the end of the surgery), 6h post-op, 12h, 24h, Day 2, Day 3, Day 7, and at any other time if necessary. The maximum pain felt is compared between the 2 groups.
Use of oral pain treatment | 7 days
  Patients reporte the consumption of analgesic treatment in a diary. The proportion of patients who took oral pain medication and the treatment categories are compared between the 2 groups.
Adverse events | 7 days
  Adverse events reported by patients on a diary from Day 0 to Day 7 and clinically observed by the dental surgeon will assess the safety and tolerability of sealers and endodontic procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Colombel, MD, Principal Investigator — Private dental practice
Locations (1):
- Cabinet dentaire, Rennes, France